CLINICAL TRIAL: NCT04646538
Title: 3 D Volume Assessment of the Periapical Healing Following Regenerative Endodontic Procedures Using Cone- Bean Computed Tomography
Brief Title: Volume Assessment of the Periapical Healing Following Regenerative Endodontic Procedures Using Cone- Bean Computed Tomography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Noha Mohamed El Kateb, lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19832009
Record Dates: First submitted 2020-11-18; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Necrotic Pulp; Periapical; Infection
Keywords: REPs; CBCT; volume; Mature teeth
MeSH Terms: conditions — Dental Pulp Necrosis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X3 group (Experimental)
  Interventions: Other: Regenerative Endodontics Procedures (REPs)

INTERVENTIONS:
Other: Regenerative Endodontics Procedures (REPs) — REPs was done for 10 mature maxillary necrotic teeth with periapical lesions. Instrumentation was done using Protaper Next system till size X3. Irrigation with 1.5 % NaOCl was done in the first visit. in the second visit, bleeding was induced in the canal by irritating the periapical area followed by the application of Biodentine as cervical plug then completion of the coronal restoration.

SUMMARY:
3D volume assessment was done to evaluate the periapical healing following REPs in mature teeth.

DETAILED DESCRIPTION:
REPs were done for 10 mature maxillary necrotic teeth with periapical lesions confirmed by digital periapical radiographs. Instrumentation was done using Protaper Next till size X3 (size 30). Pre-operative radiographs also included CBCT scans to measure the 3D volume and area of the periapical lesion to be used as baseline data. The postoperative radiographic examination included: a) digital periapical radiographs taken at 3,6,9, and 12 months to monitor the lesion through out the follow-up period. b)CBCT scan to measure quantitatively the volume and area of the periapical lesion after 12 months follow up

ELIGIBILITY:
Inclusion Criteria:

* Necrotic Mature Maxillary anterior teeth with periapical lesions.

Exclusion Criteria:

* Patients with mobile and fractured teeth

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Measurement the volume of periapical lesion preoperatively and comparing it with the new volume after REPs using cone-beam computed tomography. | 12 months
  Measuring the volume in mm3

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Kateb NME, Fata MM. Influence of periapical lesion size on healing outcome following regenerative endodontic procedures: a clinical investigation. Oral Radiol. 2022 Oct;38(4):480-489. doi: 10.1007/s11282-021-00578-8. Epub 2021 Nov 26. PMID 34826060